CLINICAL TRIAL: NCT04383691
Title: A Randomized, 6-Week, Multicenter, Double-Blind, Placebo-Controlled, Flexible Dose, Parallel-Group Study of Lurasidone for the Treatment of Bipolar I Depression
Brief Title: A Study of Lurasidone Compared With Placebo for the Treatment of Bipolar I Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company's business decision
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1071301
Record Dates: First submitted 2020-04-16; First posted 2020-05-12 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Bipolar I Depression
MeSH Terms: interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lurasidone (Experimental): Subjects will be administered orally, once daily, in the evening. Subjects will be treated with Lurasidone 20 mg/day for Days 1-2-3, 40 mg/day for Days 4-5-6, and 60 mg/day on Day 7. Flexible dosing of study drug will be permitted beginning on Day 8.
  Interventions: Drug: Lurasidone HCl
- Placebo (Placebo Comparator): Subjects will be administered orally, once daily, in the evening. Subjects will be treated with Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone HCl — Subjects will be administered orally, once daily, in the evening. Subjects will be treated with Lurasidone 20 mg/day for Days 1-2-3, 40 mg/day for Days 4-5-6, and 60 mg/day on Day 7. Flexible dosing of study drug will be permitted beginning on Day 8.
  Arms: Lurasidone
Drug: Placebo — Subjects will be administered orally, once daily, in the evening. Subjects will be treated with Placebo.
  Arms: Placebo

SUMMARY:
The study evaluates the efficacy and safety of lurasidone compared with placebo in treating Bipolar I Depression.

DETAILED DESCRIPTION:
The primary objective is to compare the efficacy of lurasidone (20-120 mg/day) monotherapy with that of placebo in patients with Bipolar I Depression by assessing the change from baseline in the MADRS total score at Week 6.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have provided written voluntary consent in person after receiving and understanding adequate explanation about the study, including the objectives, content, expected therapeutic and pharmacological effects, and risks.
2. Outpatients who are aged 18 through 65 years at time of informed consent.
3. Patients with bipolar I disorder, most recent episode depressed, without rapid cycling disease course ( no less than 4 episodes of mood disturbance in the 12 months prior to screening), and without psychotic features (diagnosed by DSM-5 criteria).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the MADRS total score at Week 6 | Baseline/ week 6
  Montgomery-Asberg Depression Rating Scale (MADRS)is a clinician-rated assessment of a subject's level of depression. The MADRS total score ranges from a minimum of 0 to a maximum of 60. For the MADRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome. The MADRS contains ten (10) items. The total score is computed as the sum of the scores for the 10 items.

SECONDARY OUTCOMES:
Change from baseline in the CGI-BP-S (depression) score at Week 6 | Baseline/ week 6
  Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) score (depression) is a clinician-rated assessment of a subject's level of depression. The CGI depression score ranges from a minimum of 1 to a maximum of 7. For the CGI depression score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.

OTHER OUTCOMES:
Change from baseline in the MADRS total score at each assessment point | Baseline/ Week 1/ Week2/ Week3/ Week4/ Week5/ Week 6
  Montgomery-Asberg Depression Rating Scale (MADRS)is a clinician-rated assessment of a subject's level of depression. The MADRS total score ranges from a minimum of 0 to a maximum of 60. For the MADRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome. The MADRS contains ten (10) items. The total score is computed as the sum of the scores for the 10 items.
Change from baseline in the CGI-BP-S (depression) score at each assessment point | Baseline/ Week 1/ Week2/ Week3/ Week4/ Week5/ Week 6
  Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) score (depression) is a clinician-rated assessment of a subject's level of depression. The CGI depression score ranges from a minimum of 1 to a maximum of 7. For the CGI depression score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
Change from baseline in the SDS total score at Week 6 | Baseline/ week 6
  Sheehan Disability Scale (SDS) total score is a subject-rated assessment of a subject's level of functional impairment in work/school, social life and family life/home responsibilities. The SDS total score ranges from a minimum of 0 to a maximum of 30. For the SDS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome. The SDS contains three (3) items. The total score is computed as the sum of the scores for the 3 items.
Change from baseline in the YMRS total score at Week 6 and each assessment point | Baseline/ Week 1/ Week2/ Week3/ Week4/ Week5/ Week 6
  YMRS (Young Mania Rating Scale) is a clinician-rated assessment of the severity of mania in subjects with a diagnosis of bipolar disorder. The YMRS total score ranges from a minimum of 0 to a maximum of 60. For the YMRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome. The YMRS contains eleven (11) items. The total score is computed as the sum of the scores for the 11 items.
Change from baseline in the HAM-A total score at Week 6 | Baseline/ week 6
  The Hamilton Rating Scale for Anxiety (HAM-A) scale is a rating scale developed to quantify the severity of anxiety symptomatology. The HAM-A total score ranges from a minimum of 0 to a maximum of 56. For the HAM-A total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome. The HAM-A contains fourteen (14) items. The total score is computed as the sum of the scores for the 14 items.
Incidence of Adverse events (AEs) and Adverse drug reactions (ADRs) | Screening/ Baseline/ Week 1/ Week2/ Week3/ Week4/ Week5/ Week 6/ Follow up
  Adverse events, adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Doctor, Principal Investigator — Beijing Anding Hospital capital medical university
Locations (26):
- China (26):
  - Beijing Anding Hospital capital medical university, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - Peking University 6th Hospital, Beijing, Beijing Municipality
  - Chongqing Mental Health Center, Chongqing, Chongqing Municipality
  - Xiamen Xianyue Hospital, Xiamen, Fujian
  - Guangzhou Huiai Hospital, Guangzhou, Guangdong
  - Shenzhen Kangning Hospital, Shenzhen, Guang
  - Hebei Provincal Mental Health Center, Baoding, Hebei
  - The 2nd Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Zhumadian Psychiatric Hospital, Zhumadian, Henan
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Brain Hospital of Hunan Province, Changsha, Hunan
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Ningbo Kangning Hospital, Ningbo, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Zhenjiang mental health center, Zhenjiang, Jiangsu
  - Dalian Seventh People's Hospital, Dalian, Liaoning
  - Jining Psychiatric prevention and treatment hospital, Jining, Shandong
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Mental Health Center of Xi'an City, Xi’an, Shanxi
  - The forth People's Hospital of Chengdu, Chengdu, Sichuan
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
  - Urumqi 4th People's Hospital, Ürümqi, Xinjiang
  - The 1st Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The 1st Hospital of Zhejiang Province, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.